# **Statistical Analysis Plan**

A Phase 3, open-label, randomized, controlled, multi-country study to evaluate the immune response, safety and reactogenicity of RSVPreF3 OA investigational vaccine when co-administered with FLU-QIV vaccine in adults aged 60 years and above.

214488

**Date of Document: 16 April 2021** 

The GlaxoSmithKline group of companies

214488 (RSV OA=ADJ-007)

**Information Type:** Statistical Analysis Plan (SAP)



## TITLE PAGE

**Protocol Title:** A Phase 3, open-label, randomized, controlled, multi-country

study to evaluate the immune response, safety and

reactogenicity of RSVPreF3 OA investigational vaccine when co-administered with FLU-QIV vaccine in adults aged 60 years

and above.

**Study Number:** 214488 (RSV OA=ADJ-007)

Compound

GSK3844766A

**Number:** 

**Abbreviated Title:** A Phase 3, open-label, randomized, controlled, multi-country

study to evaluate the immune response, safety and

reactogenicity of RSVPreF3 OA investigational vaccine when co-administered with FLU-QIV vaccine in adults aged 60 years

and above.

Sponsor Name: GlaxoSmithKline Biologicals SA (GSK)

**Regulatory Agency Identifier Number(s)** 

IND 18540 RSV PreF3 Older Adult

Registry ID

Clintrials.gov Not available

Copyright 2021 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| TIT | LE PAC | GE | 1 |
| TAE | BLE OF | CONTENTS | 2 |
| LIS | T OF T | ABLES | 4 |
| LIS | T OF F | IGURES | 5 |
| 1. | | ODUCTION | |
| | 1.1.<br>1.2. | Objectives, Estimands and Endpoints Study Design | |
| 2. | STATI | ISTICAL HYPOTHESES | 10 |
| | 2.1. | Multiplicity Adjustment | |
| 3. | ANAL' | YSIS SETS | 11 |
| | 3.1. | Criteria for eliminating data from Analysis Sets | |
| | | 3.1.1. Elimination from Exposed Set (ES) | |
| | | 3.1.2. Elimination from Per-protocol Set (PPS) | 11 |
| 4. | STATI | ISTICAL ANALYSES | 14 |
| | 4.1. | General Considerations | |
| | | 4.1.1. General Methodology | |
| | 4.0 | 4.1.2. Definitions | |
| | 4.2. | Primary Endpoint(s) Analyses | |
| | | 4.2.2. Main analytical approach | |
| | | 4.2.3. Sensitivity analyses | |
| | 4.3. | Secondary Endpoint(s) Analyses | |
| | | 4.3.1. Immunogenicity analysis | |
| | | 4.3.1.1. Between groups assessment | |
| | | 4.3.1.2. Within groups assessment | |
| | | 4.3.2. Safety analysis | |
| | 4.4. | Tertiary Analyses | |
| | | 4.4.1. Between groups assessment | |
| | 4.5. | 4.4.2. Within groups assessment | |
| | 4.5. | Safety Analyses | |
| | 4.6. | Other Analyses | |
| | 4.7. | Interim Analyses | |
| | | 4.7.1. Sequence of analyses | |
| | 4.8. | Changes to Protocol Defined Analyses | |
| 5. | SAMP | PLE SIZE DETERMINATION | 21 |
| 6. | SLIPP | PORTING DOCUMENTATION | 22 |
| <b>U</b> . | 6.1. | Appendix 1 Study Population Analyses | |
| | J. 1. | 6.1.1. Participant Disposition | |

# $214488 \mid Statistical \ Analysis \ Plan \quad 16 \ Apr \ 2021 \mid TMF-11875408 \mid 3.0$

# CONFIDENTIAL

| | | 6.1.2. | Demogra | phic and Baseline Characteristics | 23 |
|---|---|---|---|---|---|
| | | 6.1.3. | | Deviations | |
| | | 6.1.4. | | xposure | |
| | | 6.1.5. | | ant Medications | |
| | | 6.1.6. | | ant Vaccinations | |
| | | 6.1.7. | | Analyses Due to the COVID-19 Pandemic | |
| | 6.2. | Appendi | | erivations Rule | |
| | | 6.2.1. | | g events to vaccine doses | |
| | | 6.2.2. | | of missing data | |
| | | | 6.2.2.1. | Dates | |
| | | | 6.2.2.2. | Laboratory data | 25 |
| | | | 6.2.2.3. | Daily recording of solicited events | 25 |
| | | | | 6.2.2.3.1. Studies with paper diaries | |
| | | 6.2.3. | Data deriv | vation | |
| | | | 6.2.3.1. | Age at first dose in years | 26 |
| | | | 6.2.3.2. | Age category at vaccination | |
| | | | 6.2.3.3. | Temperature | |
| | | | 6.2.3.4. | Numerical serology results | |
| | | | 6.2.3.5. | Geometric mean titers (GMTs) and | |
| | | | | concentrations (GMCs) | 27 |
| | | | 6.2.3.6. | Onset day | 27 |
| | | | 6.2.3.7. | Duration of events | |
| | | | 6.2.3.8. | Counting rules for combining solicited and | |
| | | | | unsolicited adverse events | 27 |
| | | | 6.2.3.9. | Counting rules for occurrences of solicited | |
| | | | | events | 28 |
| | | | 6.2.3.10. | Counting rules for occurrence of unsolicited | |
| | | | | adverse events | 29 |
| | | 6.2.4. | Display of | f decimals | 30 |
| | | | 6.2.4.1. | Percentages | 30 |
| | | | 6.2.4.2. | Differences in percentages | |
| | | | 6.2.4.3. | Demographic/baseline characteristics statistics | |
| | | | 6.2.4.4. | Serological summary statistics | 30 |
| 7. | DEFF | DENCES | | | 20 |
| 1. | | | | | 30 |

# 214488 | Statistical Analysis Plan | 16 Apr 2021 | TMF-11875408 | 3.0

## **CONFIDENTIAL**

# **LIST OF TABLES**

| | | PAGE |
|---|---|---|
| Table 1 | List of elimination codes | 12 |
| Table 2 | Overall power to demonstrate co-primary objectives: non-<br>inferiority of the immunogenicity of RSVPreF3 OA investigational<br>vaccine when co-administered with FLU vaccine as compared to<br>when administered alone- assuming 393 participants are<br>available in each group | 22 |
| Table 3 | Evaluation of non-inferiority in terms of HI antibody SCR when the FLU vaccine is co-administered with the RSVPreF3 OA investigational vaccine as compared to FLU when administered alone assuming 393 participants are available in each group for a range of plausible SCRs. | 22 |
| Table 4 | Intensity grading scale for solicited events | 29 |

# 214488 | Statistical Analysis Plan | 16 Apr 2021 | TMF-11875408 | 3.0

# CONFIDENTIAL

# **LIST OF FIGURES**

| | | PAGE |
|----------|-----------------------|------|
| Figure 1 | Study design overview | 9 |

# **VERSION HISTORY**

| SAP<br>Version | Approval Date | Protocol Version (Date) on which SAP is Based | Change | Rationale |
|---|---|---|---|---|
| SAP | 16 Apr 2021 | 24 November 2020<br>(Protocol amendment 1) | Not<br>Applicable | Original version |

# 1. INTRODUCTION

The purpose of this SAP is to describe the planned statistical analyses for Study RSV OA=ADJ-007 (214488).

# 1.1. Objectives, Estimands and Endpoints

| Objectives | Endpoints |
|---|---|
| Co-Pri | mary |
| To demonstrate the non-inferiority of<br>RSVPreF3 OA investigational vaccine<br>when co-administered with the FLU<br>vaccine compared to RSVPreF3 OA<br>investigational vaccine administered<br>alone. | RSV-A neutralization antibody titers<br>expressed as group GMT ratio, 1<br>month after the RSVPreF3 OA<br>investigational vaccine dose. |
| To demonstrate the non-inferiority of<br>FLU vaccine when co-administered<br>with the RSVPreF3 OA<br>investigational vaccine compared to<br>FLU vaccine administered alone. | HI antibody titers for each of the FLU vaccine strains expressed as group GMT ratio, 1 month after the FLU vaccine dose. |
| Secon | dary |
| To evaluate the non-inferiority of FLU vaccine when co-administered with the RSVPreF3 OA investigational vaccine compared to FLU vaccine administered alone. | HI seroconversion status for each of<br>the FLU vaccine strains expressed as<br>SCR, 1 month after the FLU vaccine<br>dose. |
| To evaluate the humoral immune response to RSVPreF3 OA investigational vaccine when coadministered with the FLU vaccine or administered alone. | <ul> <li>RSV-A neutralization antibody titers expressed as MGI at 1 month after the RSVPreF3 OA investigational vaccine dose.</li> <li>RSV-B neutralizing antibody titers expressed as group GMT ratio and MGI at 1 month after the RSVPreF3 OA investigational vaccine dose in a subset.</li> </ul> |
| To evaluate the humoral immune response to the FLU vaccine when coadministered with the RSVPreF3 OA investigational vaccine or administered alone. | <ul> <li>HI antibody titers for each of the FLU vaccine strains expressed as GMT, at Day 1 and Day 31.</li> <li>HI seroconversion status for each of the FLU vaccine strains expressed as SCR, from Day 1 to Day 31.</li> </ul> |

| Objectives | Endpoints |
|---|---|
| | <ul> <li>HI seroprotection status for each of the FLU vaccine strains expressed as SPR, at Day 1 and Day 31.</li> <li>HI antibody titers for each of the FLU vaccine strains expressed as MGI, 1 month after the FLU vaccine dose.</li> </ul> |
| To evaluate the safety and reactogenicity following administration of the RSVPreF3 OA investigational vaccine and FLU vaccine, co-administered or administered alone. | <ul> <li>Percentage of participants reporting each solicited event with onset within 4 days after vaccine administration (i.e. the day of vaccination and 3 subsequent days).</li> <li>Percentage of participants reporting unsolicited adverse events (pIMD, non-serious AE or serious AE) within 30 days after vaccine administration (i.e. the day of vaccination and 29 subsequent days).</li> <li>Percentage of participants reporting SAEs after vaccine administration (Day 1) up to study end (6 months after last vaccination).</li> <li>Percentage of participants reporting pIMDs after vaccine administration (Day 1) up to study end (6 months after last vaccination).</li> </ul> |
| Terti | ary |
| To further evaluate the humoral immune response to RSVPreF3 OA investigational vaccine when coadministered with the FLU vaccine or administered alone. | RSVPreF3-specific IgG concentrations expressed as group GMC ratio and MGI at 1 month after the RSVPreF3 OA investigational vaccine dose in a subset. |

FLU vaccine is referring to FLU-QIV; IgG: Immunoglobulin G; GMT: Geometric Mean Titer; GMC: Geometric Mean Concentration; HI: Hemagglutinin Inhibition; pIMD: potential immune-mediated disease. AE: adverse event; SAE: serious adverse event.

SCR: Seroconversion rate: the percentage of vaccinees who have either a HI pre-dose titer < 1:10 and a post-dose titer ≥ 1:40 or a pre-dose titer ≥ 1:10 and at least a four-fold increase in post-dose titer.

SPR: Seroprotection rate: The percentage of vaccinees with a serum HI titer ≥ 1:40 that usually is accepted as indicating protection.

MGI: The geometric mean of the within participant ratios of the post-dose titer over the pre-dose titer.

#### **Primary estimand**

The primary clinical question of interest is to show non inferiority of the RSVPreF3 OA investigational vaccine and the FLU vaccine when co-administered versus separate administration 1 month apart in eligible participants who complied with the study requirements as defined per protocol (refer to section 3 for the definition of the per protocol set used for the primary analysis and to section 4.2.2 for the statistical method).

# 1.2. Study Design

The current study is designed to assess the immunogenicity, safety and reactogenicity of the RSVPreF3 OA investigational vaccine when co-administered with a FLU vaccine, compared with administration of the vaccines separately. There are 2 parallel arms:

- **Co-Ad group:** Participants will receive a single dose of RSVPreF3 OA investigational vaccine and a single dose of FLU vaccine at Visit 1 (Day 1).
- **Control group**: Participants will receive a single dose of FLU vaccine at Visit 1 (Day 1), followed by a single dose of the RSVPreF3 OA investigational vaccine at Visit 2 (Day 31).

All participants will be followed up for safety for 6 months after the last study vaccine administration.

Randomization (1:1) Co-Ad group Control group N≈440 VISIT 1 VISIT 3 VISIT 2 Visits/ Day 1 Day 31 Day 61 CONTACT Baseline for Co-Ad group 1MPD for Co-Ad group 1MPD for FLU No visit for Co-Ad group 1MPD for RSV in Control Contact 6 months post-last and for FLU in Control group **Timepoints** dose = Baseline for RSV in Control group group FLU+RSV (Co-Ad) 🧪 🧳 Vaccination FLU 🥖 RSV 🥖 Sample BS BS BS\* collection Safety Solicited events up to 4 days post-dose monitoring Unsolicited AEs up to 30 days post-dose All SAEs and pIMDs up to study end Study end SAEs related to study participation or to a concurrent GSK medication/vaccine up to study end AEs/SAEs leading to withdrawal from the study up to study end

Figure 1 Study design overview

1MPD = 1 month post-dose.

Testing of RSV-B neutralizing antibodies and RSVPreF3 IgG will be performed on a random subset of participants (approximately 220 participants each from the Co-Ad group and the Control group).

<sup>\*</sup> Blood sample only from participants in Control group.

FLU = FLU-QIV; RSV = RSVPreF3 OA investigational vaccine; BS = Blood sample from all participants (except for blood sample at Visit 3 which is only applicable for Control group).

Note: Unsolicited AEs will be collected from first dose to 30 days post-dose. SAEs and pIMDs will be collected from first dose through the entire study period. SAEs related to study participation will be collected from the time of consent.

## 2. STATISTICAL HYPOTHESES

The study includes 2 confirmatory co-primary objectives.

• To demonstrate the non-inferiority of RSVPreF3 OA investigational vaccine when co-administered with the FLU vaccine compared to RSVPreF3 OA investigational vaccine administered alone in terms of RSV-A neutralization antibody GMT ratio at 1 month after the RSVPreF3 OA investigational vaccine dose (i.e. at Day 31(Visit 2) for the Co-Ad group and at Day 61(Visit 3) for the Control group).

# Null hypothesis vs. Alternative hypothesis:

 $H_0: \mu_{Control\ group}/\mu\ _{Co\text{-Ad\ group}} \geq log(1.5)\ vs.\ H_a: \ \mu_{Control\ group}/\ \mu\ _{Co\text{-Ad\ group}} \leq log(1.5)$ 

where  $\mu$  represents the expected mean of log transformed RSV-A neutralization antibody titers at 1 month after the RSVPreF3 OA investigational vaccine dose. The null hypothesis will be rejected if the upper limit of the two-sided 95% CI for the group GMT ratio (Control group divided by Co-Ad group) in RSV-A neutralization antibody titers 1 month after the RSVPreF3 OA investigational vaccine dose  $\leq$  1.5.

• To demonstrate the non-inferiority of FLU vaccine when co-administered with the RSVPreF3 OA investigational vaccine compared to FLU vaccine administered alone in terms of HI GMT ratio for each of the FLU vaccine strains at 1 month after the FLU vaccine (i.e. at Day 31(Visit 2) for both groups).

### **Null hypothesis vs. Alternative hypothesis:**

 $H_0\text{: }\mu_{Control\ group}/\mu\ \text{Co-Ad\ group} \geq log(1.5)\ vs.\ H_a\text{: }\mu_{Control\ group}/\mu\ \text{Co-Ad\ group} \leq log(1.5)$ 

where  $\mu$  represents the expected mean of log transformed HI antibody titers at 1 month after the FLU vaccine dose. The null hypothesis will be rejected if the upper limit of the two-sided 95% CI for the group GMT ratio (Control group divided by Co-Ad group) in HI antibody titers for each of the FLU vaccine strains 1 month after the FLU vaccine  $\leq 1.5$ .

# 2.1. Multiplicity Adjustment

The success of the study depends on the success of all co-primary objectives. Using a nominal alpha of 2.5% for each of them will ensure the global type I error for the co-primary objectives is controlled below 2.5%.

### 3. ANALYSIS SETS

| Analysis Set | Definition / Criteria |
|---|---|
| Enrolled set | Participants who agreed to participate in a clinical study after completion of the informed |
| | consent process*. |
| Safety/Exposed | All participants who received a study intervention. Analysis per group is based on the study |
| set (ES) | intervention administered. |
| Per-Protocol set | All eligible participants who received at least one study intervention as per protocol, had |
| (PPS) immunogenicity results pre-post-dose for at least one antigen, complied with blood draw | |
| | intervals (refer to intervals mentioned below) and contribution of participants to PPS at specific |
| | timepoint will be defined by timepoint, without intercurrent medical conditions that may interfere |
| | with immunogenicity and without prohibited concomitant medication/vaccination. |

<sup>\*</sup>All participants enrolled and included in the database will be part of the enrolled set.

Intervals for the Co-Ad group: Visit1-Visit2=30-42 days

Intervals for the Control group: Visit1-Visit2=30-42 days, Visit2-Visit3=30-42 days

# 3.1. Criteria for eliminating data from Analysis Sets

Elimination codes will be used to identify participants to be eliminated from analysis. Detail is provided below for each set.

# 3.1.1. Elimination from Exposed Set (ES)

Code 1010 (Vaccine number not allocated),1030 (Study intervention not administered at all), 800 (Fraudulent data) and code 900 (invalid informed consent) will be used for identifying participants eliminated from ES (see Table 1).

# 3.1.2. Elimination from Per-protocol Set (PPS)

A participant will be excluded from the populations for analysis under the following conditions:

- For codes 800, 900, 1030, 1050 and 2020: participants will be eliminated for all visits.
- For codes 1040, 1070, 1080, 1090, 2010, 2040, 2050, 2080: participants will be eliminated from a specific visit (at which the condition is met) onwards.
- For codes 2090, 2100, 2120: participants will be eliminated at the specific visit at which the condition is met. RSV-B neutralizing antibody titers and RSVPreF3-specific IgG concentrations are tested only in a subset of participants.

Table 1 List of elimination codes

| Code | Condition under which the code is used | Visit<br>/Contact(timepoints)<br>where the code is<br>checked | Visit from when it is applicable | Applicable for analysis set/endpoint |
|---|---|---|---|---|
| 800 | Fraudulent data | All | All | ES and PPS<br>for analysis of<br>immunogenicity |
| 900 | Invalid informed consent | All | All | ES and PPS<br>for analysis of<br>immunogenicity |
| 1030 | Study intervention not administered at all | All | All | ES and PPS<br>for analysis of<br>immunogenicity |
| 1040 | Administration of concomitant vaccine(s) forbidden in the protocol Use of any investigational or non- registered vaccine other than the study interventions during the period beginning 30 days before the first dose of study vaccines and ending 30 days after the last vaccine administration, or planned use during the study period. Planned or actual administration of a vaccine not foreseen by the study protocol in the period starting 30 days before the first study intervention administration and ending 30 days after the last study intervention administration. Note: In case an emergency mass vaccination for an unforeseen public health threat (e.g.: a pandemic) is recommended and/or organized by the public health authorities, outside the routine immunization program, the time period described above can be reduced if necessary for that vaccine provided it is used according to the local governmental recommendations and that the Sponsor is notified accordingly. | Visit 1,2,3 | From the specific visit the condition is met | PPS for analysis of immunogenicity |
| 1050 | Randomisation failure: Subject not randomized in the correct group (To be attributed by Statistician only; Check SBIR, replacement, vaccine administration) | Visit 1 | All | PPS for<br>analysis of<br>immunogenicity |
| 1070 | Vaccine administration not according to protocol Incomplete vaccination course Participant was vaccinated with the correct vaccine but containing a lower volume Wrong replacement or study vaccine administered (not compatible with the vaccine regimen associated to the treatment number) Route of the study vaccine is not intramuscular | Vaccination visit(s) 1<br>or 1 and 2 as<br>applicable | From the specific visit (1 or 2) the condition is met as applicable for the respective group | PPS for<br>analysis of<br>immunogenicity |

| Code | Condition under which the code is used | Visit /Contact(timepoints) where the code is checked | Visit from when it is applicable | Applicable for analysis set/endpoint |
|---|---|---|---|---|
| | Side of administration wrong (for Co-ad group if both vaccines are given in the same arm) Wrong reconstitution of administered vaccine | | | |
| 1080 | Vaccine temperature deviation Vaccine administered despite a Good Manufacturing Practices (GMP) no-go temperature deviation | Vaccination visit(s) 1 or 1 and 2 as applicable | From the specific visit (1 or 2) the condition is met as applicable for the respective group | PPS for<br>analysis of<br>immunogenicity |
| 1090 | Expired vaccine administered | Vaccination visit(s) 1<br>or 1 and 2 as<br>applicable | From the specific visit (1 or 2) the condition is met as applicable for the respective group | PPS for<br>analysis of<br>immunogenicity |
| 2010 | Protocol violation linked to inclusion/exclusion criteria All inclusion/exclusion criteria defined in the protocol to be checked. | Visit 1,2,3 | From the specific visit (1,2 or 3) the condition is met. | PPS for analysis of immunogenicity |
| 2020 | All Pre-dose results are missing:<br>RSV-A and HI for the FLU vaccine strains | Co-Ad group: Visit 1<br>Control group: Visit 1<br>and Visit 2 | All | PPS for analysis of immunogenicity |
| 2040 | Administration of any medication forbidden by the protocol Use of any investigational or non- registered drug, or medical device other than the study interventions during the period beginning 30 days before the first dose of study vaccines and ending 30 days after the last vaccine administration, or planned use during the study period. Administration of long-acting immune- modifying drugs or planned administration at any time during the study period (e.g. infliximab). Administration of immunoglobulins and/or any blood products or plasma derivatives planned administration during the study period. Chronic administration (defined as more than 14 consecutive days in total) of immunosuppressants or other immune- modifying drugs planned administration during the study period. For corticosteroids, this will mean prednisone ≥20 mg/day, or equivalent. Inhaled and topical steroids are allowed. | Visit 1,2,3 | From the specific visit (1,2 or 3) the condition is met | PPS for analysis of immunogenicity |
| 2050 | Intercurrent medical condition: Participants may be eliminated from the PPS for immunogenicity if, during the study, they incur a condition that has the | Visit 1,2,3 | From the specific visit (1,2 or 3) the condition is met | PPS for analysis of immunogenicity |

| Code | Condition under which the code is used | Visit /Contact(timepoints) where the code is checked | Visit from when it is applicable | Applicable for analysis set/endpoint |
|---|---|---|---|---|
| | capability of altering their immune response (intercurrent medical condition) or are confirmed to have an alteration of their initial immune status. | | | |
| 2080 | Participants did not comply with vaccination schedule for the control group number of days between dose 1 and dose 2 is outside [30-42 days] | Visit 2 | Visit 3 for the control group | PPS for analysis of immunogenicity |
| 2090 | Participants did not comply with blood sample schedule: Co-Ad group: Number of days between vaccination (visit1) and blood sample (visit2) is outside [30-42] days Control group: Number of days between vaccination (visit1) and blood sample (visit2) or (visit2) and blood sample (visit3) is outside [30-42] days | Visit 2, Visit 3 as applicable for the group | At the specific visit (2 or 3) the condition is met as applicable for the respective group | PPS for analysis of immunogenicity |
| 2100 | Serological results not available at the post dose time point for all antigens tested at that particular time point. | Visit 2,3 | At the specific visit (2 or 3) the condition is met as applicable for the respective group | |
| 2120 | Obvious incoherence/abnormality or error in laboratory data Unreliable released data as a result of confirmed sample mismatch or confirmed inappropriate sample handling at lab | Visit 2, Visit 3 | At the specific visit (2 or 3) the condition is met as applicable for the respective group | PPS for<br>analysis of<br>immunogenicity |

### 4. STATISTICAL ANALYSES

### 4.1. General Considerations

## 4.1.1. General Methodology

95% CI for proportion will be based on exact Clopper-Pearson confidence interval.

95% CI for group difference in proportion will be based on Miettinen and Nurminen confidence interval.

The group GMT ratio will be based on a back transformation of group contrast in an ANCOVA model applied to the logarithm- transformed titers. The ANCOVA model will include the treatment group, the age category (age at vaccination: 60-69, 70-79 or ≥80 years), country and sex as fixed effects and the pre-dose log-10 titer as regressors.

95% CI for GMT will be based on a back transformation of student CI for the mean of log-transformation.

### 4.1.2. Definitions

• For the RSV antigens:

A seronegative participant will be defined as a participant whose antibody titer/concentration is below the cut-off value of the assay. A seropositive participant is a participant whose antibody titer/concentration is greater than or equal to the cut-off value of the assay.

MGI (mean geometric increase): The geometric mean of the within participant ratios of the post-dose titer over the pre-dose titer.

• For the FLU antigens:

SCR (seroconversion rate): The percentage of vaccinees who have either a HI predose titer < 1:10 and a post-dose titer  $\ge 1:40$  or a pre-dose titer  $\ge 1:10$  and at least a four-fold increase in post-dose titer.

HI SPR (seroprotection rate): The percentage of vaccinees with a serum HI titer  $\geq$ 1:40 that usually is accepted as indicating protection.

MGI (mean geometric increase): The geometric mean of the within participant ratios of the post-dose titer over the pre-dose titer.

# 4.2. Primary Endpoint(s) Analyses

The primary analysis will be based on the PPS for analysis of immunogenicity. If, in any vaccine group, the percentage of vaccinated participants with serological results excluded from the PPS for analysis of immunogenicity is 5% or more, a second analysis based on the ES will be performed to complement the PPS analysis.

## 4.2.1. Between groups assessment

- The 2-sided 95% CI for the group GMT ratio in terms of RSV-A neutralizing antibody titers between RSVPreF3 OA investigational vaccine administered alone (Control group) over RSVPreF3 OA investigational vaccine when co-administered with the FLU vaccine (Co-Ad group) will be computed at 1 month after the RSVPreF3 OA investigational vaccine dose (i.e. at Day 31(Visit 2) for the Co-Ad group and at Day 61(Visit 3) for the Control group).
- The 2-sided 95% CI for the group GMT ratio in terms of HI antibody titers for each of the FLU vaccine strains between RSVPreF3 OA investigational vaccine administered alone (Control group) over RSVPreF3 OA investigational vaccine when co-administered with the FLU vaccine (Co-Ad group) will be computed at 1 month after the FLU vaccine (i.e. at Day 31 (Visit 2) for both groups):

## 4.2.2. Main analytical approach

The 2-sided 95% CI for group GMT ratio will be derived from an ANCOVA model\* on log<sub>10</sub> transformed titer.

\*The model will include the treatment group, the age category (age at vaccination: 60-69, 70-79 or ≥80 years), country and sex as fixed effects, and the pre-dose log10-transformed titer as covariate. Missing data will not be replaced. Titers below the assay cut-off will be replaced by half the assay cut-off, titers above the upper-limit of quantification (ULOQ) will be replaced by the ULOQ.

Success criteria for non-inferiority:

- 1. The upper limit of the 2-sided 95% CI on the group GMT ratio (Control group divided by Co-Ad group) for RSV investigational vaccine is ≤1.5.
  - AND
- 2. The upper limit of the 2-sided 95% CI on the group GMT ratio (Control group divided by Co-Ad group) for each of the FLU vaccine strains are ≤1.5.

# 4.2.3. Sensitivity analyses

Not applicable.

# 4.3. Secondary Endpoint(s) Analyses

# 4.3.1. Immunogenicity analysis

The primary analysis of secondary immunogenicity endpoints will be based on the PPS for analysis of immunogenicity. If, in any vaccine group, the percentage of vaccinated participants with serological results excluded from the PPS for analysis of immunogenicity is 5% or more, a second analysis based on the ES will be performed to complement the PPS analysis.

#### 4.3.1.1. Between groups assessment

- The asymptotic standardized 95% CI for the difference in seroconversion rate (Control group minus Co-Ad group) will be computed at 1 month after the FLU vaccine (i.e. at Day 31 (Visit 2) for both groups).
  - Reference criteria for evaluation of non-inferiority:
  - The upper limit of the 2-sided 95% CI on the group difference (Control group minus Co-Ad group) in seroconversion rate is  $\leq$ 10% for anti-HI antibodies.
- The 2-sided 95% CI for the group GMT ratio in terms of RSV-B neutralizing antibody titers between RSVPreF3 OA investigational vaccine administered alone (Control group) over RSVPreF3 OA investigational vaccine when co-administered with the FLU vaccine (Co-Ad group) will be computed at 1 month after the RSVPreF3 OA investigational vaccine dose (i.e. at Day 31 (Visit 2) for the Co-Ad group and at Day 61 (Visit 3) for the Control group) in a subset of participants.
  - All between groups analyses of secondary endpoints presented in this section will be descriptive with the aim to characterize the difference in immunogenicity between groups. These descriptive analyses should be interpreted with caution considering that there is no adjustment for multiplicity for these comparisons.

### 4.3.1.2. Within groups assessment

For each group, at each time point that blood samples are collected for humoral immune response and for each assay (unless otherwise specified):

- Percentage of participants above pre-defined assay cut-off and their exact 95% CI will be tabulated.
- Percentage of participants above seroprotection/seroconversion rate for HI antibody titer and their exact 95% CI will be tabulated.
- Percentage of participants above seroprotection/seroconversion rate by age group (60-64 YOA, ≥65 YOA) for HI antibody titer and their exact 95% CI will be tabulated.
- GMCs/GMTs and their 95% CI will be tabulated.
- MGI will be tabulated with 95% CI.
- Antibody titer/concentration will be displayed using reverse cumulative curves.
   The analysis of RSV-B neutralizing antibodies will be performed in a subset of participants.
  - The above mentioned descriptive within group immunogenicity analysis will also be generated by age at first vaccination (60-69, 70-79,  $\geq$  65,  $\geq$  70 and  $\geq$ 80 years).
- Additionally, the CBER and CHMP criteria for HI SPR and SCR will be assessed as follows:

CBER criteria to be evaluated:

- The lower limit (LL) of the 95% CI for SCR should be ≥40% in participants aged 18-64\* YOA or ≥30% in participants ≥65 YOA.
- The LL of the 95% CI for SPR should be ≥70% in participants aged 18-64\*
   YOA or ≥60% in participants ≥65 YOA.
  - \*In this study, only participants from 60 YOA and higher are included, hence we can expect only a small proportion of participants in this category of 60 to 64 years. Although the SCR will be estimated the criteria cannot be evaluated for this category.

### CHMP criteria to be evaluated:

- At least one of the 3 following criteria should be met:
- the point estimates of SPR >60%, SCR >30%, and MGI >2.0 for elderly > 60 years for each of the antigen strains.

These above defined analyses evaluating the CBER and CHMP criteria should be interpreted with caution considering that there is no adjustment for multiplicity for these comparisons.

### 4.3.2. Safety analysis

The safety analysis will be performed on the ES as follows:

- The number and percentage of participants and doses with at least one administration site event AE (solicited and unsolicited), with at least one systemic AE (solicited and unsolicited) and with any AE during the 4-day and 30-day follow-up period will be tabulated with exact 95% confidence interval (CI) after each dose and overall. The same computations will be done for Grade 3 AEs, for Grade 3 non-serious AEs and for AEs resulting in a medically attended visit.
  - These analyses will present all solicited and unsolicited AEs, including SAEs and pIMDs (unless otherwise specified).
  - The above analysis will also be performed for the solicited symptoms only during the 4-day follow-up period.
- The number and percentage of participants reporting each individual solicited administration site AE (any grade, Grade 3 and resulting in medically attended visit) and solicited systemic AE (any grade, Grade 3 and resulting in medically attended visit) during the 4-day follow-up period (i.e. the day of vaccination and 3 subsequent days) will be tabulated for each group after each dose and overall. The percentage of doses followed by each individual solicited administration site AE (any grade, Grade 3 and resulting in medically attended visit) and solicited systemic AE (any grade, Grade 3 and resulting in medically attended visit) during the 4-day follow-up period (i.e. the day of vaccination and 3 subsequent days) will be tabulated, with exact 95% CI.
- For fever, the number and percentage of participants reporting fever by half degree (°C) cumulative increments during the 4-day follow-up period (i.e. the day of vaccination and 3 subsequent days) will be tabulated for each group after each dose and overall.
- The percentage of participants with each solicited administration site event and solicited systemic event (any grade and grade 3) will be represented graphically for each group after each dose.
- The number of days with solicited events reported during the 4-day follow-up period will be tabulated for each individual solicited event using descriptive statistics (mean, minimum, Q1, median, Q3, maximum). The same computations will be done for Grade 3 solicited events.
- The number and percentage of participants with any unsolicited AEs during the 30-day follow-up period (i.e. the day of vaccination and 29 subsequent days) with its exact 95% CI will be tabulated by group and by Medical Dictionary for Regulatory Activities (MedDRA) preferred term. Similar tabulation will be done for Grade 3 unsolicited AEs, for any causally related unsolicited AEs, for Grade 3 causally related unsolicited AEs and for unsolicited AEs resulting in a medically attended visit. The verbatim reports of unsolicited AEs will be reviewed by a physician and the signs and symptoms will be coded according to the MedDRA Dictionary for Adverse Reaction Terminology. Every verbatim term will be matched with the appropriate Preferred Term. The above analysis by dose will also be performed.

- The number and percentage of participants with at least one report of SAE classified by the MedDRA Preferred Terms and reported after vaccine administration (Day 1) up to study end (6 months after last vaccination) will be tabulated with exact 95% CI.
- The number and percentage of participants with at least one report of causally related SAE classified by the MedDRA Preferred Terms and reported after vaccine administration (Day 1) up to study end (6 months after last vaccination) will be tabulated with exact 95% CI.
- The same tabulation will be presented for fatal SAEs.
- All SAEs will also be described in detail in a tabular listing.
- All pIMD will also be described in detail in a tabular listing.
- All AEs/SAEs leading to study/intervention discontinuation from dose 1 up to study end will be tabulated.
- The percentage of participants with at least one report of pIMD classified by the MedDRA Preferred Terms and reported after vaccine administration (Day 1) up to study end (6 months after last vaccination) will be tabulated with exact 95% CI. The percentage of participants with at least one report of related pIMD classified by the MedDRA Preferred Terms and reported after vaccine administration (Day 1) up to study end (6 months after last vaccination) will be tabulated with exact 95% CI.
- The number and percentage of participants using concomitant medication (any medication and any antipyretic) during the 4-day and the 30-day follow-up period after each dose and overall will be tabulated with exact 95% CI.
- Compliance in completing solicited events information will be tabulated after each dose and overall.
- Some of the key safety analysis will be generated by age group at first vaccination  $(60-69, 70-79, \ge 65, \ge 70 \text{ and } \ge 80 \text{ years})$  as mentioned below.
  - The number and percentage of participants reporting each individual solicited administration site AE (any grade, Grade 3 and resulting in medically attended visit) and solicited systemic AE (any grade, Grade 3 and resulting in medically attended visit) during the 4-day follow-up period (i.e. the day of vaccination and 3 subsequent days) will be tabulated for each group after each dose and overall.
  - The number and percentage of participants with any unsolicited AEs during the 30-day follow-up period (i.e. the day of vaccination and 29 subsequent days) with its exact 95% CI will be tabulated by group and by Medical Dictionary for Regulatory Activities (MedDRA) preferred term.
- For clinicaltrials.gov and EudraCT posting purposes, percentage of participants of combined solicited and unsolicited non-serious adverse events during the 30-day follow-up period (i.e. the day of vaccination and 29 subsequent days) will be produced by System Organ Class and preferred terms and according to occurrence of each event.

## 4.4. Tertiary Analyses

The below analysis will be performed on the PPS for analysis of immunogenicity for the RSVPreF3 IgG ELISA concentration in a subset of participants.

## 4.4.1. Between groups assessment

- The 2-sided 95% CI for the group GMT ratio in terms of RSVPreF3 IgG ELISA concentration between RSVPreF3 OA investigational vaccine administered alone (Control group) over RSVPreF3 OA investigational vaccine when co-administered with the FLU vaccine (Co-Ad group) will be computed at 1 month after the RSVPreF3 OA investigational vaccine dose (i.e. at Day 31 for the Co-Ad group and at Day 61 for the Control group)
- The above defined between groups analysis will be descriptive with the aim to characterize the difference in immunogenicity between groups. These descriptive analyses should be interpreted with caution considering that there is no adjustment for multiplicity of this comparison.

## 4.4.2. Within groups assessment

For each group, at each time point that blood samples are collected for humoral immune response, the below analysis will be performed:

- Percentage of participants above pre-defined assay cut-off and their exact 95% CI will be tabulated.
- GMCs and their 95% CI will be tabulated.
- MGI will be tabulated with 95% CI.
- Antibody titer/concentration will be displayed using reverse cumulative curves.

# 4.5. Safety Analyses

Safety analyses are described in Section 4.3.2.

#### 4.5.1. COVID-19 Assessment and COVID-19 AEs

A standardized MedDRA Query (SMQ) will be used to identify all COVID-19 AEs.

The overall incidence of COVID-19 AEs and SAEs , COVID-19 AEs leading to study intervention discontinuation, COVID-19 AEs leading to study withdrawal, and severe COVID-19 AEs will be summarized. The incidence of these events at individual PT level can be obtained from the standard AE/SAE summaries.

COVID-19 assessments (confirmed, probable and suspected diagnosis) for participants with COVID-19 AEs will be summarized.

The number and percentage of participants with concomitant vaccination (COVID-19) before and during the study will be tabulated with exact 95% CI.

# 4.6. Other Analyses

Not Applicable.

# 4.7. Interim Analyses

There are no interim analyses planned for this study.

# 4.7.1. Sequence of analyses

A final analysis will be conducted once all the immunogenicity data are available for primary and secondary endpoints. This final analysis will include immunogenicity and safety data up to Visit 2 (Co-Ad group) or Visit 3 (Control group).

An EoS analysis with all data including the data obtained until 6 months post-last dose will be performed.

# 4.8. Changes to Protocol Defined Analyses

Change from the defined analysis set specified in the protocol amendment 1 (Dated: 24 November 2020) are detailed below.

| Protocol Defined Analysis set | SAP Defined Analysis set | Rationale for Change |
|---|---|---|
| All eligible participants who received all study intervention as per protocol, had immunogenicity results pre-post-dose for at least one antigen, complied with blood draw intervals (refer to Table 3 of protocol) and contribution of participants to PPS at specific timepoint will be defined by timepoint, without intercurrent medical conditions that may interfere with immunogenicity and without prohibited concomitant medication/vaccination. | All eligible participants who received at least one study intervention as per protocol, had immunogenicity results pre-post-dose for at least one antigen, complied with blood draw intervals (refer to intervals mentioned below) and contribution of participants to PPS at specific timepoint will be defined by timepoint, without intercurrent medical conditions that may interfere with immunogenicity and without prohibited concomitant medication/vaccination. | It is appropriate to include the participant in the analysis of Flu even if the RSV vaccine was not administered |

### 5. SAMPLE SIZE DETERMINATION

The target enrolment will be 880 participants (440 in the group receiving the RSVPreF3 OA investigational vaccine co-administered with the FLU vaccine (Co-Ad group) and 440 in the Control group where RSVPreF3 OA investigational vaccine and FLU vaccine are administered staggered) to obtain at least 786 evaluable participants (393 in the Co-Ad group and 393 in Control group) for the evaluation of the primary objectives, assuming that approximately 10% of the enrolled participants will not be evaluable.

Each objective will be evaluated with a nominal type I error of 2.5%.

Table 2 Overall power to demonstrate co-primary objectives: non-inferiority of the immunogenicity of RSVPreF3 OA investigational vaccine when co-administered with FLU vaccine as compared to when administered alone- assuming 393 participants are available in each group

| RSV Non-inferiority* (1-sided test with alpha = 2.5%) | | | | |
|---|---|---|---|---|
| Endpoint | Standard deviation of log10 concentration | Non-<br>inferiority<br>margin | Type II error | Power |
| GMTs RSV-A neutralization antibody | 0.45 | 1.5 | 0.02% | 99.98% |
| FLU Non-inferiority* (1-sided test with alpha = 2.5%) | | | | |
| Endpoint | Standard deviation of log10 concentration | Non-<br>inferiority<br>margin | Type II error | Power |
| GMTs HI H1N1 strain | 0.6 | 1.5 | 1.58% | 98.42% |
| GMTs HI H3N2 strain | 0.6 | 1.5 | 1.58% | 98.42% |
| GMTs HI B/Washington strain | 0.6 | 1.5 | 1.58% | 98.42% |
| GMTs HI B/Phuket strain | 0.6 | 1.5 | 1.58% | 98.42% |
| Global Type II error to show non-infer | | | | |
| Global power | ~93.7% | | | |

<sup>\*</sup>Pass 2019 alpha = 2.5%, Two-Sample T-Tests for Non-Inferiority Assuming Equal Variance and Equal mean.

Considering identical true GMTs in both groups with a common population standard error of 0.45 for the RSV-A neutralization antigen and 0.6 for each of the FLU strains in log10 transformed concentration, the study has at least 93.7% power to meet the coprimary objectives.

#### Nominal powers to evaluate secondary objective

The nominal power to evaluate the non-inferiority on seroconversion rate for each of the FLU strains is above 79%, depending on the plausible rates.

Table 3 Evaluation of non-inferiority in terms of HI antibody SCR when the FLU vaccine is co-administered with the RSVPreF3 OA investigational vaccine as compared to FLU when administered alone assuming 393 participants are available in each group for a range of plausible SCRs

| N evaluable participants per group | Threshold | Plausible rates in Control group** | Type II<br>error# | Nominal Power |
|---|---|---|---|---|
| | | FLU vaccine: Non-inferiority* in terms of SCR | | |
| 393 | 10% | 70% | 13.4% | 86.6% |
| 393 | 10% | 50% | 20.4% | 79.6% |
| 393 | 10% | 35% | 16.1% | 83.9% |
| 393 | 10% | 25% | 10.1% | 89.9% |

SCR: Seroconversion Rate.

<sup>\*</sup>Pass 2019 alpha = 2.5%, for SCR – Non-inferiority: Proportions – Two independent Proportions – Non-Inferiority Tests for the Difference Between Two Proportions based on Miettinen and Nurminen method

<sup>\*\*</sup> SCR observed in the Control group in Zoster-004 study range from 35.3% to 60.9%.

<sup>\*</sup>The overall power for this secondary objective will be 100-sum of the type II error for each of the 4 strains.

## 6. SUPPORTING DOCUMENTATION

# 6.1. Appendix 1 Study Population Analyses

### 6.1.1. Participant Disposition

The number of participants who withdraw from the study will be tabulated by group according to the reason for drop-out. This analysis will be based on the ES and the PPS.

## 6.1.2. Demographic and Baseline Characteristics

The median, mean, range and standard deviation of age (in years) at first vaccination will be computed by group. The center distribution, distribution of participants in each age category (60-69, 70-79,  $\geq$  65,  $\geq$  70 and  $\geq$ 80 years), geographical ancestry and sex composition will be presented. This analysis will be based on the ES and the PPS.

Medical history will be summarized respectively.

#### 6.1.3. Protocol Deviations

The number of participants enrolled into the study as well as the number of participants excluded from per protocol set (PPS) analyses will be tabulated for the total population. This analysis, also broken down by study group, will be based on the ES.

The number of participants enrolled into the study as well as the number of participants excluded from per the ES will be tabulated for the total population. This will be based on all enrolled participants.

## 6.1.4. Subject exposure

The number and percentage of participants who received the co-administered vaccine and the control vaccine will be tabulated by group and by vaccine for the ES.

#### 6.1.5. Concomitant Medications

The number and percentage of participants and doses using concomitant medication (any medication, any antipyretic and any antipyretic taken prophylactically, respectively) during the 4-day follow-up period (i.e., on the day of vaccination and 3 subsequent days) and during the 30-day follow-up period (i.e., on the day of vaccination and 29 subsequent days) will be summarized by group after each vaccine dose and overall

### 6.1.6. Concomitant Vaccinations

Not applicable.

### 6.1.7. Additional Analyses Due to the COVID-19 Pandemic

Depending on how the Covid-19 situation evolves, the SAP might be amended to reflect the analysis corresponding to Covid-19."

# 6.2. Appendix 2 Data Derivations Rule

This section contains standard rules for data display and derivation for clinical and epidemiological studies.

## 6.2.1. Attributing events to vaccine doses

The dose relative to an event is the most recent study dose given to a participant prior to the start of a given event. For example, if the start date of an adverse event is between Dose 1 and Dose 2, the relative dose will be Dose 1.

If an event starts on the same day as a study dose, the relative dose will be derived from the additional information provided in the case report form (CRF) using the contents of the flag indicating if the event occurred before or after study dose. If 'after study dose' is selected, the relative dose for the event will be the one administered on the start day of the event. If 'before study dose' is selected, the relative dose for the event will be the dose prior to this one.

### 6.2.2. Handling of missing data

#### 6.2.2.1. Dates

When partially completed dates (i.e. dates missing a day and/or month) are used in calculations, the following standard rules will be applied:

- A missing day will be replaced by 15
- A missing day and month will be replaced by June 30<sup>th</sup>.

The following exceptions apply:

When partially completed dates (i.e. with missing day or month) are used in calculations, the following rules will be applied:

- Adverse event start dates with missing day:
  - If the month is not the same as the vaccine dose, then the imputed start date will be the 1<sup>st</sup> of the month
  - If the event starts in the same month as the vaccine dose, the flag indicating if the event occurred before or after vaccination (AE.AESTRTPT) will be used to complete the date. If 'after vaccination' is selected, the imputed start date will match the vaccine dose given during that month. If 'before vaccination' is selected, the imputed date will be one day before the vaccine dose given during that month.
- Adverse event start dates with missing day and month:
  - If the year is not the same as the vaccine dose, then the imputed start date will be the 1<sup>st</sup> of January.

- If the event starts in the same year as the vaccine dose, the flag indicating if the event occurred before or after vaccination (AE.AESTRTPT) will be used to complete the date. If 'after vaccination' is selected, the imputed start date will match the first vaccine dose given during that year. If 'before vaccination' is selected, the imputed date will be one day before the first vaccine dose given during that year.
- Adverse event end dates with missing day: the imputed end date will be the last day of the month (30 or 31) or the study conclusion date whichever comes first.
- Adverse event end dates with missing day and month: the imputed end date will be the last day of the year (31st of December) or the study conclusion date whichever comes first.

All incomplete concomitant medication/vaccination start/end date will follow the rules above.

### 6.2.2.2. Laboratory data

Missing laboratory results (including immunological data) will not be replaced.

### 6.2.2.3. Daily recording of solicited events

## 6.2.2.3.1. Studies with paper diaries

For studies using paper diaries which have questions in the CRF indicating the presence or absence of solicited events, the following rules are applicable:

- Denominators for the summary of administration site (or systemic) solicited events will be calculated using the number of participants who respond "Yes" or "No" to the question concerning the occurrence of administration site (or systemic) events.
- When a specific solicited event is marked as having not occurred following a specific study dose (i.e. SDTM CE.CEOCCUR=N for the specified post-dose period for the event in question), all daily measurements will be imputed as Grade 0.
- When a specific solicited event is marked as having occurred following a specific study dose (i.e. SDTM CE.CEOCCUR=Y for the specified post-dose period for the event in question), any missing daily recordings will be given imputed values to allow them to contribute to the 'Any' rows but not to specific grade rows of the solicited event summary tables.
- When the occurrence of a specific solicited event is not present (i.e. SDTM CE.CEOCCUR is neither Y nor N for the specified post-dose period for the event in question) but the group of solicited events (administration site or systemic) is marked as having occurred (i.e. SDTM CE.CEOCCUR=Y), all missing daily recordings will be given imputed values to allow them to contribute to the 'Any' rows but not to specific grade rows of the solicited event summary tables.

The following table shows how participants contribute to each category for a specific solicited event over the Day X to Day Y post-dose period:

| Solicited event category | Participants included in the calculation of the numerator |
|---|---|
| Any | All participants with at least one occurrence of the adverse event at grade 1, grade 2, or grade 3 between Day X and Day Y or with the adverse event marked as present and at least one missing daily recording between Day X and Day Y |
| At least grade 1 | All participants with at least one occurrence of the adverse event at grade 1, grade 2, or grade 3 between Day X and Day Y |
| At least grade 2 | All participants with at least one occurrence of the adverse event at grade 2 or grade 3 between Day X and Day Y |
| At least grade 3 | All participants with at least one occurrence of the adverse event at grade 3 between Day X and Day Y |

## 6.2.3. Data derivation

### 6.2.3.1. Age at first dose in years

Age will be calculated as the number of years between the date of birth and the date of first vaccination.

In case of partial dates, the following 2 dates will be used as replacement dates:

- 15th of month, if the day is missing.
- 30th of June, if day and months are missing.

### 6.2.3.2. Age category at vaccination

As only the year of birth will be collected in the eCRF, there might be some discrepancies between the age computed using standard derivation rules and the age category used in SBIR for the minimization.

Therefore, for the analysis by age, the age categories will be determined according to the information entered in SBIR (add name of variable in SDTM), except for "≥65 YOA" category which will be obtained using the derived age because this category is not used in SBIR for minimization.

## 6.2.3.3. Temperature

Temperatures will be presented in degrees Celsius (°C). Temperatures reported in degrees Fahrenheit (°F) will be converted as follows:

Temperature (Celsius) =  $((Temperature (Fahrenheit) - 32) \times 5)/9$ 

### 6.2.3.4. Numerical serology results

Numerical serology results will be derived from the content of IS.ISORRES in the SDTM dataset. For assays with a specific cut-off, the following derivation rules apply:

| IS.ISORRES | Derived value |
|-----------------------------------------|---------------|
| "NEG", "-", or "(-)" | cut-off/2 |
| "POS", "+", or "(+)" | cut-off |
| "< value" and value is <= assay cut-off | cut-off/2 |
| "< value" and value is > assay cut-off | value |
| "> value" and value is < assay cut-off | cut-off/2 |
| "> value" and value is >= assay cut-off | value |
| "value" and value is < cut-off | cut-off/2 |
| "value" and value is >= cut-off | Value |
| "value" and value is > ULOQ | ULOQ |
| All other cases | missing |

### 6.2.3.5. Geometric mean titers (GMTs) and concentrations (GMCs)

Geometric Mean Titer (GMT) or Concentration (GMC) calculations are performed by taking the inverse logarithm of the mean of the log titer or concentration transformations. Non quantifiable antibody titers or concentrations will be converted as described in section 6.2.3.4 for the purpose of GMT/GMC calculation. Cut-off values are defined by the laboratory before the analysis.

#### 6.2.3.6. Onset day

The onset day for an event (e.g. AE, concomitant medication/vaccination) is the number of days between the last study dose and the start date of the event. This is 1 for an event occurring on the same day as a study dose (and reported as starting after study dose).

#### 6.2.3.7. Duration of events

The duration of an event with a start and end date will be the difference between the start and end date plus one day, i.e. an event that starts on 3 March 2018 and ends on 12 March 2018 has a duration of 10 days.

The duration of solicited events will be calculated as the sum of the individual days with the adverse event reported at grade 1 or higher during the solicited event period.

### 6.2.3.8. Counting rules for combining solicited and unsolicited adverse events

For output combining solicited and unsolicited adverse events, all serious adverse events will be considered systemic events since the administration site flag is not included in the expedited adverse event CRF pages. Unsolicited adverse events with missing administration site flag will also be considered systemic.

Solicited events will be coded by MedDRA as per the following codes:

| Solicited event | Lower level term code | Corresponding Lower level term decode |
|---|---|---|
| Pain | 10022086 | Injection site pain |
| Erythema | 10015150 | Erythema |
| Swelling | 10053425 | Injection site swelling |
| Fever | 10016558 | Pyrexia |
| Headache | 10019211 | Headache |
| Fatigue | 10016256 | Fatigue |
| Myalgia | 10028411 | Myalgia |
| Arthralgia | 10003239 | Arthralgia |

The latest available MedDRA version will be used for coding

Multiple events with the same preferred term which start on the same day are counted as only one occurrence.

### 6.2.3.9. Counting rules for occurrences of solicited events

When the occurrences of solicited events are summarized, each event recorded as having occurred during a specific period will be counted as only one occurrence regardless of the number of days on which it occurs. Also, in the case of co-administered study interventions, an administration site event recorded for a participant following multiple study interventions will be counted as only one occurrence.

### Table 4 Intensity grading scale for solicited events



The maximum intensity of local injection site erythema/swelling and fever will be scored at GSK as follows:

CCI - This section contained Clinical Outcome Assessment data collection questionnaires or ndices, which are protected by third party copyright laws and therefore have been excluded.

### 6.2.3.10. Counting rules for occurrence of unsolicited adverse events

Unsolicited adverse event summaries are including serious adverse events unless specified otherwise.

As per CDISC Vaccines Therapeutic Area guide, the solicited events which continue beyond the observation period are stored in the Adverse Events (AE) domain but they do not contribute to the summaries of unsolicited adverse events.

Missing severity, relationship with study vaccine, and outcome of unsolicited adverse events will not be replaced and will appear as 'UNKNOWN' when displayed in a statistical output.

### 6.2.4. Display of decimals

## 6.2.4.1. Percentages

Percentages and their corresponding confidence limits will be displayed with one decimal except for 100% in which case no decimal will be displayed.

### 6.2.4.2. Differences in percentages

Differences in percentages and their corresponding confidence limits will be displayed with two decimals.

### 6.2.4.3. Demographic/baseline characteristics statistics

The mean, median, and standard deviation for continuous baseline characteristics (height, weight, body mass index (BMI), pre-dose body temperature) will be presented with one decimal.

The minimum and maximum values and quartile values (if required) will be presented with the same number of decimals as the observed values.

The maximum and minimum of transformed body temperatures will be displayed with one decimal.

### 6.2.4.4. Serological summary statistics

For each assay, geometric mean titers (GMT) or concentrations (GMC) and their confidence limits will be presented with one decimal, as well as GMT/GMC fold increase from pre-dose.

GMT or GMC group ratios and their confidence limits will be displayed with 2 decimals regardless of the actual values.

#### 7. REFERENCES

Clopper CJ, Pearson E. The Use of Confidence or Fiducial Limits Illustrated in the case of the Binomial. *Biometrika*. 1934;26:404-13.

Miettinen, O. S. and Nurminen, M. Comparative analysis of two rates. Statistics in Medicine, 1985;4,213-226.